CLINICAL TRIAL: NCT07185802
Title: Clinical Outcome of Intra Articular Injection of Autologous Platelet Rich Plasma in Anterior Cruciate Ligament Injury.
Acronym: ACL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Isfath Fauzia, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5744
Record Dates: First submitted 2025-09-19; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament
Keywords: PRP in ACL injury
MeSH Terms: interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A/Experimental group (Experimental): Will receive PRP and conventional conservative method (physical therapy, functional bracing, lifestyle modification)
  Interventions: Biological: PRP injection; Other: conventional conservative method (physical therapy, functional bracing, lifestyle modification)
- Group B/Control group (Active Comparator): Will receive conventional conservative method (physical therapy, functional bracing, lifestyle modification) only
  Interventions: Other: conventional conservative method (physical therapy, functional bracing, lifestyle modification)

INTERVENTIONS:
Biological: PRP injection — Ultrasound guided intraarticular PRP is given to the patient with partial ACL tear
  Other Names: PRP group
  Arms: Group A/Experimental group
Other: conventional conservative method (physical therapy, functional bracing, lifestyle modification) — conventional conservative method (physical therapy, functional bracing, lifestyle modification)
  Other Names: Rehabilitation

SUMMARY:
This clinical trial will evaluate the effectiveness of platelet-rich plasma (PRP) injections for patients with anterior cruciate ligament (ACL) injury. ACL injuries commonly cause knee instability, pain, and reduced function, and rehabilitation alone may not fully restore recovery in all patients. PRP is prepared from a small sample of the patient's own blood and contains natural growth factors that may promote healing and improve joint function.

In this study, participants will be randomly assigned to one of two groups. The experimental group will receive a single ultrasound-guided injection of PRP into the knee joint along with a standard rehabilitation program. The control group will receive the rehabilitation program alone.

Participants will be followed up at 3 weeks, 8 weeks, and 16 weeks after treatment. At each follow-up visit, knee function, pain level, and physical performance will be assessed using validated outcome measures. The primary aim is to determine whether PRP provides additional benefit compared with rehabilitation alone in improving function and reducing symptoms in ACL-injured patients.

This study will provide new evidence about the role of PRP in ACL management, which may help guide future treatment decisions.

ELIGIBILITY:
Inclusion criteria:

* Patients of both sexes who are older than 18 years and younger than 50 years
* 3 or Less than 3-months history of knee injuries
* ACL injury MRI Grade 1 (Low) and medium Grade 2 (Medium) grade
* ACL injury associated with Grade 1 or 2 Posterior cruciate ligament (PCL) tear and/or Grade 1 or 2 meniscal tear
* The Complete Blood Count (CBC) report shows a hemoglobin > 10gm/dl and platelet count >150,000/microliter prior to the procedure
* Capable of comprehending informed consent

Exclusion criteria:

* Patients who have had intra articular corticosteroid injections in the index knee during the last 12 weeks
* Patients who are taking systemic steroid
* Patients who are younger than 18 and older than 50 years
* Those with a history of platelet disorders or on the therapeutic anticoagulant or anti platelet drugs
* Hemoglobin below 10 gm/dl
* Platelet count <150000/microliter
* Complete tear of both bundles on MRI
* Grade 3 or more PCL and meniscal tear on MRI
* Previous or concurrent ligament reconstruction in the index knee joint.
* Connective tissue disorders like Marfan Syndrome, Ehler-Danlos Syndrome etc.
* Any inflammatory disease like Rheumatoid Arthritis, spondyloarthritis, gout, pseudogout etc involving the knee joint.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS ): Change in pain intensity measured by Visual Analog Scale | Baseline, 3 weeks, 8 weeks, and 16 weeks after intervention.
  Pain intensity will be assessed using the Visual Analog Scale (0 = no pain, 10 = worst possible pain).

SECONDARY OUTCOMES:
KOOS: Change in functional outcome measured by Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 3 weeks, 8 weeks, and 16 weeks after intervention.
  KOOS assesses five domains: pain, symptoms, activities of daily living, sport/recreation function, and knee-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Isfath Fauzia, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh; Prof. Dr. Md. Ali Emran, MBBS, FCPS, Study Chair — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh; Dr. Md. Nuruzzaman Khandaker, MBBS, FCPS, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh; Dr. Md. Tariqul Islam, MBBS, FCPS, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
I will think later in case of mind change